CLINICAL TRIAL: NCT02219880
Title: Kava for the Treatment of Generalised Anxiety Disorder: A Double-Blind Randomised Placebo-Controlled Trial
Acronym: KGAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Swinburne University of Technology (Other); The University of Queensland (Other)
Responsible Party: Principal Investigator, Jerome Sarris, Dr Jerome Sarris, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 137/14
Record Dates: First submitted 2014-08-13; First posted 2014-08-19 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Generalized Anxiety Disorder
Keywords: Kava; Anxiety; Generalized Anxiety Disorder; Psychiatric; Anxiolytic; GABA; Kavalactones
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Inert tablets matched for colour, size and consistency to active arm treatment. Both treatment arm tablets will match in appearance, and neither participants nor the trial clinicians will know what they are taking.
  Interventions: Dietary Supplement: Placebo
- Kava - standardised 240mg kavalactones (Experimental): Standardised 240mg kavalactones per day - fixed dose regime of two tablets of kava twice per day
  Interventions: Dietary Supplement: Kava (240mg of kavalactones per day)

INTERVENTIONS:
Dietary Supplement: Kava (240mg of kavalactones per day) — Kava 60 milligrams per tablet = 240mg of kavalactones per day
  Other Names: Kava; Kavalactones; Piper methysticum
  Arms: Kava - standardised 240mg kavalactones
Dietary Supplement: Placebo — Inert tablets containing vegetable fibre matched for colour, size and consistency to active arm treatment.
  Arms: Placebo

SUMMARY:
The use of Kava in Generalised Anxiety Disorder: an 18-week double-blind, randomised, placebo-controlled study.

DETAILED DESCRIPTION:
The primary aim is to confirm the efficacy and safety of Kava compared to placebo in Generalized Anxiety Disorder (GAD). Secondary aims of the study are to confirm the relationship between specific genetic variations and response to Kava, and to explore the effects of Kava on the expression of specific genes.

Consenting participants will be randomly allocated to take either Kava or placebo over 18 weeks. They will be assessed at regular interviews throughout the trial and will have four blood tests (liver function tests to monitor participant safety, and collection of genetic material providing information on neurochemistry). The design of the study is a multi-centre, 18-week, 2-arm, double-blind randomised clinical trial (RCT) using a standardised pharmaceutical-grade water-soluble extract of Kava (240mg of kavalactones per day) versus placebo in 210 adults with GAD.

ELIGIBILITY:
To be considered for inclusion in this study, participants will be required to meet the following criteria:

* Aged between 18-70 years
* Meets the Diagnostic and Statistical Manual (DSM) IV and DSM-V diagnostic criteria for generalised anxiety disorder (GAD) based on structured interview (Mini International Neuropsychiatric Interview-Plus 6 [MINI-Plus 6]. Note that while the MINI-Plus 6 uses the DSM-IV criteria, the same criteria are used in the DSM-V).
* Presents with anxiety (Hamilton Anxiety Rating Scale ≥ 18) at the time of study entry
* Fluent in written and spoken English
* Provides a signed copy of the consent form

Participants are ineligible to enter the trial if they have any of the following conditions:

* Primary diagnosis other than GAD
* Presentation of moderate to severe depressive symptoms (Montgomery-Asberg Rating Scale: MADRS ≥ 18 at time of study entry or ≥ 24 at any time during study)
* Presentation of suicidal ideation (≥ 3 on MADRS suicidal thoughts domain at time of study entry or at any time during study)
* Current diagnosis of bipolar disorder or schizophrenia on structured interview (MINI Plus)
* Current substance/alcohol use disorder on structured interview (MINI Plus) Page 21 of 39 Commercial-in-Confidence
* Currently taking an antidepressant, mood stabiliser, antipsychotic, anticonvulsant, warfarin or thyroxin, or current regular use (more than 2 days per week) of a benzodiazepine or opioid-based analgesic
* Current use of a psychotropic nutraceutical (e.g. St John's wort)
* Previous intolerance to kava
* Three or more failed trials of pharmacotherapy for the current GAD episode
* Recently commenced psychotherapy (within four weeks of study entry)
* Known or suspected clinically unstable systemic medical disorder
* Diagnosed hepato-biliary disease/inflammation
* Elevated liver enzymes at baseline blood test
* Pregnancy or breastfeeding, or trying to conceive
* Not using medically approved contraception (including abstinence) if female and of childbearing age
* Unable to participate in all scheduled visits, treatment plan, or other trial procedures according to the protocol (except for the optional genetic component)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAMA) - change in score | 18 weeks
  Reduction of participant's anxiety will be assessed on the HAMA from baseline to week 16 across time used a mixed methods model.

SECONDARY OUTCOMES:
Gamma-aminobutyric acid (GABA) transporter polymorphisms moderating response to study intervention | 18 weeks
  Will assess whether response to Kava will be moderated by gamma-aminobutyric acid (GABA) transporter polymorphisms. Specifically, whether rs2601126-T allele or rs2697153-A allele carriers have greater reduction of anxiety

OTHER OUTCOMES:
Changes in score to psychometric questionnaire measures | 18 weeks
  Depressive symptoms on the Montgomery-Asberg Depression Rating Scale (MADRS), self-rated anxiety on the Beck Anxiety Inventory (BAI), pathological worry on the Penn State Worry Questionnaire (PSWQ), and health-related quality of life on the Short Form Survey-12 (SF-12) will also be significantly improved by Kava over placebo; and
Monoamine and GABA differential gene expression | 8 weeks
  Differential gene expression will be assessed from baseline to week 8 from participants in the Melbourne site. This will determine whether Kava increases expression of genes effecting expression of neurochemical e.g. GABA, and monoamines

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Sarris, PhD, Principal Investigator — The University of Melbourne and The Melbourne Clinic
Locations (2):
- Australia (2):
  - Royal Brisbane & Women's Hospital, Brisbane, Queensland
  - Centre for Human Psychopharmacology - Swinburne University, Melbourne, Victoria

REFERENCES:
- [Derived] Savage K, Sarris J, Hughes M, Bousman CA, Rossell S, Scholey A, Stough C, Suo C. Neuroimaging Insights: Kava's (Piper methysticum) Effect on Dorsal Anterior Cingulate Cortex GABA in Generalized Anxiety Disorder. Nutrients. 2023 Oct 28;15(21):4586. doi: 10.3390/nu15214586. PMID 37960239
- [Derived] Sarris J, Byrne GJ, Bousman CA, Cribb L, Savage KM, Holmes O, Murphy J, Macdonald P, Short A, Nazareth S, Jennings E, Thomas SR, Ogden E, Chamoli S, Scholey A, Stough C. Kava for generalised anxiety disorder: A 16-week double-blind, randomised, placebo-controlled study. Aust N Z J Psychiatry. 2020 Mar;54(3):288-297. doi: 10.1177/0004867419891246. Epub 2019 Dec 8. PMID 31813230
- [Derived] Savage KM, Stough CK, Byrne GJ, Scholey A, Bousman C, Murphy J, Macdonald P, Suo C, Hughes M, Thomas S, Teschke R, Xing C, Sarris J. Kava for the treatment of generalised anxiety disorder (K-GAD): study protocol for a randomised controlled trial. Trials. 2015 Nov 2;16:493. doi: 10.1186/s13063-015-0986-5. PMID 26527536